CLINICAL TRIAL: NCT02426164
Title: Analgesic Efficacy of Liposomal Bupivacaine in Total Knee Arthroplasty
Brief Title: Liposomal Bupivacaine in Total Knee Arthroplasty
Status: Withdrawn | Phase: Phase 4 | Type: Interventional
Why Stopped: Could not receive facility approval
Sponsor: Miller Orthopedic Specialists (Other)
Collaborators: Creighton University Medical Center (Other); CHI Health Mercy Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 633913
Record Dates: First submitted 2015-04-14; First posted 2015-04-24 (Estimated); Last update posted 2016-03-22 (Estimated); Status verified 2015-04

CONDITIONS: Pain, Postoperative; Arthroplasty, Replacement, Knee; Osteoarthritis
MeSH Terms: conditions — Pain, Postoperative; Osteoarthritis | interventions — Bupivacaine; Morphine; Epinephrine; Methylprednisolone

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Liposomal bupivacaine (Active Comparator): Periarticular infiltration of 20cc of liposomal bupivacaine with 20cc of normal saline administered prior to cementation of knee implants
  Interventions: Drug: Liposomal bupivacaine
- bupivacaine HCl, morphine, epinephrine, methylprednisolone (Active Comparator): Periarticular infiltration of 24c of bupivacaine HCl, 0.8cc morphine, 0.3cc epinephrine, and 1cc of methylprednisolone administered prior to cementation of knee implants
  Interventions: Drug: bupivacaine HCl, morphine, epinephrine, methylprednisolone

INTERVENTIONS:
Drug: Liposomal bupivacaine — Periarticular infiltration of the liposomal bupivacaine with 20cc of normal saline
  Other Names: Exparel
  Arms: Liposomal bupivacaine
Drug: bupivacaine HCl, morphine, epinephrine, methylprednisolone — Periarticular infiltration of 24c of bupivacaine HCl, 0.8cc morphine, 0.3cc epinephrine, and 1cc of methylprednisolone
  Arms: bupivacaine HCl, morphine, epinephrine, methylprednisolone

SUMMARY:
Liposomal bupivacaine is a novel local anesthetic designed for prolonged pain relief. Despite its long-acting analgesic potential, liposomal bupivacaine is significantly more expensive than other local anesthetic alternatives. The primary aim of this investigation is to examine whether or not liposomal bupivacaine provides superior pain relief or clinically significant opioid-sparing effects versus a control to justify its cost.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing a primary unilateral total knee arthroplasty by the PI of the trial

Exclusion Criteria:

* Patients with a sensitivity to marcaine
* Pregnant or lactating women
* Non-English speaking individuals

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-06; Primary Completion 2017-06 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Mean visual analog scale (VAS) pain scores | Night of surgery
  Self-reported pain scores from 0=no pain to 10=severe pain
Mean visual analog scale (VAS) pain scores | Post-operative day 1
  Self-reported pain scores from 0=no pain to 10=severe pain
Mean visual analog scale (VAS) pain scores | Post-operative day 2
  Self-reported pain scores from 0=no pain to 10=severe pain
Pain assessment phone call | Post-operative day 3
  Subjects will be called on post-operative day three by one of the investigators of the study. Subjects will be asked to rate their current pain level from 1 to 10 and to rate their worst pain level from 1 to 10 that day.

SECONDARY OUTCOMES:
Complications | Complications will be followed for the duration of patients' hospital stay, an expected average of 2-3 days.
  Number of patients with complications

CONTACTS AND LOCATIONS:
Overall Officials: Clifford K Boese, MD, Principal Investigator — Miller Orthopedic Specialists
Locations (1):
- Miller Orthopedic Specialists, Council Bluffs, Iowa, United States